CLINICAL TRIAL: NCT05742529
Title: Cosmotic Outcome of Distal Penile Hypospidias Repair Using Stitch by Stitch Glanuloplasty Versus TIP ; a Non Randamized Retrospective Study
Brief Title: Cosmotic Outcome of Distal Penile Hypospidias Repair Using Stitch by Stitch Glanuloplasty Versus TIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Tomas Mokhtar Shafik, resident of urololgy department sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: soh-Med-23-01-23
Record Dates: First submitted 2023-02-12; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Distal Penile Hypospadias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIP (Active Comparator)
  Interventions: Procedure: TIP
- stitch by stitch (Active Comparator)
  Interventions: Procedure: STITCH BY STITCH

INTERVENTIONS:
Procedure: TIP — TIP An 8F straight sound is passed into the hypospadiac meatus to assess skin coverage over the urethra., a circumscribing incision is made 2 mm proximal to the meatus, a U-shaped incision is extended proximally to healthy skin The key step in the operation is a midline relaxing incision made from within the meatus to the distal extent of the plate. This incision extends through the epithelial surface of the plate deeply into underlying connective tissues down to the corpora cavernosaNext, a 6F stent is passed into the bladder for postoperative urinary diversion. Then the urethral plate is tubularized. , stitches are ever taken further distally to ensure the neomeatus has a generous oval openingticular closures. .
  Arms: TIP
Procedure: STITCH BY STITCH — SBS in brief Operative technique :starts with penile degloving, preparation of the flap (Site of hypospadic meatus is determined after degloving). Creation of a narrow strip of the urethral plate with wide glanular wings is done using bilateral incisions which are extended to the tip of the glans. The width of the urethral plate is about 3 mm then we suture the flap to the narrow urethral plate in two layers in continuous manner using vicryl 6/0 over a suitable plastic catheter. Triangular (Vshape) area of the distal part of the flap is excised a the midline. After this we anastomose the flap to thetip of the glans. The glans appears opened in the midline as inverted V shape. Closure of the glans is finished in the midline using three mattress interrupted sutures with another three simple stitches are used in between
  Arms: stitch by stitch

SUMMARY:
Hypospadias is generally defined as the combination of three anatomic anomalies of penis, which are an abnormal ventral opening of the urethral orifice, ventral curvature of the penis, and abnormal distribution of the foreskin around the glans with a ventrally deficient hooded foreskin . It is estimated that about 1 in every 200 babies is born with hypospadias in the United States, making it one of the most common birth defects.

In newborn males, hypospadias is the second most common congenital anomaly after undescended testis. Due to incomplete closure of the penile structures during embryogenesis, the urethral opening is displaced along the ventral side of the penis . Most hypospadias occur as an isolated condition, but associated anomalies include uni/bilateral cryptorchidism and micropenis .

Duckett proposed the most commonly used classification; i.e., nearly 70% of hypospadias are either glanular or distally located on the penis and are considered a mild form, whereas the remainder is more severe and complex The main goal for hypospadias repair is to achieve both cosmetic and functional normality. Reasons for treating hypospadias include spraying of urinary stream, inability to urinate in standing position, curvature leading to difficulties during intercourse, fertility issues because of difficulty with sperm deposition, and decreased satisfaction with genital appearance. Current guidelines consider optimal age for hypospadias repair somewhere between 6 and 18 months, depending on the severity and the need for multiple procedures .

Penile biometrical parameters, like a small glans width and narrow urethral plate, are some of the anatomical factors associated with increased postoperative complications and form a technical challenge . Functional outcome was considered satisfactory when the patient could micturate an ideal stream of urine (single, compact, rifled, non-dispersed urinary stream of adequate caliber) without straining. Cosmetic outcome was considered satisfactory when a straight penis was obtained with a vertical slit like, wide, smooth external meatus at the tip of a conical glans .

The normal meatus is a vertical slit with smooth and sharp edges that is centrally located within the glans penis . The literature lacks standardization of techniques for hypospadias repair and uniform definitions of complications and outcome assessment .

Many surgical techniques have been described for glans closure and meatoplasty with variable outcomes, but none of them fits all patients with hypospadias; each procedure has its limitations and demands specific selection criteria.

Duckett described the "meatal advancement and glanuloplasty incorporated" (MAGPI) procedure. The two essential elements of MAGPI are meatoplasty and glanuloplasty. However, many researchers reported a high incidence of partial meatal regression in their patients following the MAGPI procedure.

In 1928, Mathieu described a single-stage, meatal based flap technique to repair the distal forms of hypospadias but results in flat meatus. In 2000 Boddy and Samuel reported the "V-incision" sutured MAVIS technique to provide a cosmetically acceptable natural slit-like meatus in Mathieu cases Rich et al. in 1989 described a urethral plate incision (hinging) as a modification of the Mathieu repair to improve the cosmetic outcome of the neo-meatus. It helps in achieving a slit-like vertical meatus. Nevertheless, a healthy wide urethral plate with no scarring is essential for a successful outcome Snodgrass extended the concept of urethral plate hinging by incising the whole urethral plate in the midline from the hypospadias meatus distally. It helps in the tabularization of the plate with a good cosmetic outcome.

-stitch by stitch technique: Operative technique :starts with penile degloving, preparation of the flap (Site of hypospadic meatus is determined after degloving). Creation of a narrow strip of the urethral plate with wide glanular wings is done using bilateral incisions which are extended to the tip of the glans. The width of the urethral plate is about 3 mm then we suture the flap to the narrow urethral plate in two layers in continuous manner using vicryl 6/0 over a suitable plastic catheter. Triangular (Vshape) area of the distal part of the flap is excised a the midline. After this we anastomose the flap to thetip of the glans. The glans appears opened in the midline as inverted V shape. Closure of the glans is finished in the midline using three mattress interrupted sutures with another three simple stitches are used in between

ELIGIBILITY:
Inclusion Criteria:

* Age: 1 year - 3 years old.
* Type of hyposidas: Distal penile hypospadias
* Urethral plate: if urethral plate is more than 8 mm the child was selected for TIP procedure & if the urethral plate was less than 8 mm the child was selected for stitch by stich technique

Exclusion Criteria:

* - Age: less than 1 year & more than 3 years old.
* Proximal penile hypospadias
* Previous hypospadias repair
* Raised serum creatinine, coagulopathy

Ages: 1 Year to 3 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
meatal position | 24 months
  meatal position to be at the tip of penis according to HOPE SCORE BY ( other pediatric surgeon nurse parents)
meatal shape | 24 months
  meatal shape to be vertical slit within the glans penis according to HOPE SCORE BY (other pediatric surgeon nurse parents
shape of glans | 24 months
  to be conical in shape according to HOPE SCORE BY (other pediatric surgeon nurse parents

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kojima Y, Kohri K, Hayashi Y. Genetic pathway of external genitalia formation and molecular etiology of hypospadias. J Pediatr Urol. 2010 Aug;6(4):346-54. doi: 10.1016/j.jpurol.2009.11.007. Epub 2009 Dec 7. PMID 19995686
- [Background] Bouty A, Ayers KL, Pask A, Heloury Y, Sinclair AH. The Genetic and Environmental Factors Underlying Hypospadias. Sex Dev. 2015;9(5):239-259. doi: 10.1159/000441988. Epub 2015 Nov 28. PMID 26613581
- [Background] Hsieh MH, Breyer BN, Eisenberg ML, Baskin LS. Associations among hypospadias, cryptorchidism, anogenital distance, and endocrine disruption. Curr Urol Rep. 2008 Mar;9(2):137-42. doi: 10.1007/s11934-008-0025-0. PMID 18419998
- [Background] Duckett JW Jr. Hypospadias. Pediatr Rev. 1989 Aug;11(2):37-42. doi: 10.1542/pir.11-2-37. No abstract available. PMID 2668910